CLINICAL TRIAL: NCT01309191
Title: Microarray Analysis of Scalp Biopsies in Subjects With Androgenetic Alopecia Before and After the Use of Topical Minoxidil
Brief Title: Microarray Analysis of Scalp Biopsies After Minoxidil Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: University of California, San Francisco (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 12-10-24; 338259 (Other Grant/Funding Number: Johnson & Johnson)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic Alopecia; Minoxidil; Microarray
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minoxidil (Experimental): Patients received Minoxidil (same strength as sold over the counter) twice a day for 8 weeks.
  Interventions: Other: Minoxidil
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Minoxidil — Over the counter Rogaine, twice a day for 8 weeks
  Other Names: Rogaine
  Arms: Minoxidil
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Minoxidil treatment affects hair growth in patients with male pattern baldness or androgenetic alopecia.

DETAILED DESCRIPTION:
The most common type of hair loss is androgenetic alopecia (AGA), also known as male pattern balding, or hereditary thinning. In AGA, there is a gradual transformation of large terminal hair follicles to miniaturized ones under the influence of circulating androgens that produce smaller and finer hairs with a shorter anagen cycle. This transformation, which can be seen as early as the prepubescent years, occurs only in certain regions of the scalp: the frontal hairline, top and vertex scalp. The temporo-occipital region is largely unaffected even in those with extensive balding.

The first drug to be approved for the FDA for the treatment of AGA was topical minoxidil solution (TMS). Despite its successful use, the mechanism of action of TMS is not well understood. Minoxidil is a potent vasodilator and potassium channel opener, but its mechanism of action in promoting hair regrowth appears to be independent of its vasodilation properties. Improved knowledge of the changes in gene expression associated with AGA before and after treatment with TMS and compared to placebo may lead to a greater understanding of the underlying mechanisms of action of TMS. Furthermore, there is potential for identification of those patients who would best respond to or benefit from treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male
2. Is in general good health
3. Has a diagnosis of androgenic alopecia with hair loss in both the vertex and the frontal area, Hamilton (as modified by Norwood) Type IV-V
4. Has read, signed and received a copy of the Informed Consent Form prior to initiation of the study procedures
5. Is willing to follow all instructions and able to participate in the entire study, returning for all specified visits
6. Between the age of 18 to 49 years old, inclusively

Exclusion Criteria:

1. Evidence of concomitant skin diseases of the scalp including but not limited to dandruff, seborrheic dermatitis, psoriasis, lichenoid eruption, tinea capitis or other scalp infections or infestations.
2. Has a history of recurring dandruff symptoms or seborrheic dermatitis, evidence of excoriations, or other history that might indicate an inability to use the products supplied for the duration of the study.
3. Has consistently used any medicated shampoos or anti-dandruff shampoo treatment products over the past year or at all during the two months prior to the Baseline visit.
4. Has a history of alopecia areata, totalis, universalis or any other hair loss disorder except male pattern baldness.
5. Evidence of significant scalp scarring.
6. Has skin cancer or actinic keratoses currently within the balding area.
7. Has a history of skin cancer on the scalp.
8. Has undergone a hair transplant or scalp reduction surgery.
9. Has exhibited hypersensitivity, rash or other abnormal skin reactions, symptoms or lesions to topically applied hair care products in the past year.
10. Has been diagnosed with hypothyroidism or hyperthyroidism within the past year.
11. Has taken or applied any of the following medications known to induce hypotrichosis (abnormal hair loss), and/or hypertrichosis (abnormal hair growth).

    Medications taken or used in the past 6 months
    * Finasteride -hair growth product (PropeciaÒ or ProscarÒ)
    * Topical or systemic hair growth products (commercial or investigative) e.g. minoxidil (RogaineÒ), NioxinÒ, dutasteride
    * Chemotherapeutic agents
    * Systemic Retinoids (e.g. acitretin, etretinate, isotretinoin, Vitamin A > 5,000 IU (per day)
    * Immunosuppressives (e.g. tacrolimus, cyclosporine A)
    * Antimetabolic agents. (e.g. FludaraÒ, LeustatinÒ
    * Antimitotic agents
    * Anti-androgens (e.g. flutamide, spironolactone, cyproterone acetate)
    * Androgens (e.g. testosterone, methyl testosterone, danazol)
    * DHEA, androstenedione
    * Ketaconazole -systemic (antifungal)
    * Ginseng (herb)
    * Saw Palmetto
    * Diazoxide (hyperglycemic, antihypertensive agent)
    * Anticoagulants (e.g. dicumarol, heparin, warfarin)
    * Interferon
    * Beta blockers (e.g. AcebutololÒ,, AtenololÒ, propranolol, TimololÒ, MetoprololÒ)
    * Antiepileptic and anticonvulsants (e.g. valproic acid, carbamazepine, diphenylhydantoin)
    * Antithyroid drugs (e.g. carbimazole, methimazole, methylthiouracil, propylthiouracil)
    * Topical corticosteroids on scalp or applied to more than 25% of the body surface area
    * Systemic corticosteroids
    * Topical ketaconazole shampoo or cream
12. Has a significant medical condition including, but not limited to:

    Hypertension (acceptable if controlled by other than a beta blocker); angina, myocardial infarction; history of fainting or dizziness; history of kidney or urinary disorders; diabetes; hemophilia or any condition determined by the Investigator as significant and therefore considered a cause for exclusion
13. Has recently been on, or is currently on a medically managed weight reduction program.
14. Has had a significant febrile illness (high fever lasting several days) within 8 weeks of the Baseline visit.
15. Has participated in an investigational drug study within 4 weeks of the Baseline visit.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Analysis of change in gene expression before and after topical minoxidil application | at baseline and after 8 weeks of treatment
Differences ing ene expression in two different regions of the scalp, frontal and vertex. | Baseline and after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pratima Karnik, Ph.D., Principal Investigator — UH Case Medical Center
Locations (1):
- Skin Study Center, UH Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Price VH. Treatment of hair loss. N Engl J Med. 1999 Sep 23;341(13):964-73. doi: 10.1056/NEJM199909233411307. No abstract available. PMID 10498493